CLINICAL TRIAL: NCT00398125
Title: A Phase 2a, Multicenter, Randomized, Parallel, Double-Blind, Dose Ranging, Placebo-Controlled Study to Compare Antiviral Effect, Safety, Tolerability and Pharmacokinetics of GSK364735 Monotherapy Versus Placebo Over 10 Days in HIV-1 Infected Adults.
Brief Title: Monotherapy Versus Placebo Over 10 Days in Integrase Naive HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRZ107460
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV-1 Infection
Keywords: GSK364735; HIV-1; integrase inhibitor
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — GSK364735

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK364735

SUMMARY:
To investigate safety, tolerability and anti-viral activity in Integrase-Naïve HIV-1 infected adults

ELIGIBILITY:
Inclusion criteria:

* Documented HIV-1 infection with screening viral load between 5000 and 300,000 copies/mL.
* Baseline CD4 cell count greater than 100.
* Females must be of non-childbearing potential
* Not have received antiretroviral therapy in the 12 weeks prior to first dose.

Exclusion criteria:

* Must not be infected with hepatitis B or C.
* Patients must not have any acute laboratory abnormality.
* Must not have any active CDC (Centers for Disease Control and Prevention)Category C disease (1993), except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in viral load | from Day 1 to Day 11
Amount of drug in blood | on Days 1 and 10.

SECONDARY OUTCOMES:
Immunologic effect Development of resistance mutations Viral load change and drug levels in semen for a group of patients | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Dallas, Texas